CLINICAL TRIAL: NCT02868996
Title: An Open Label, Phase 1b, Single CENTER, Ascending Dose Study TO ASSESS THE SAFETY AND TOLERABILITY of DM199 With a Comparative Pharmacokinetic Study of DM199 Administered Intravenously and a Bioavailability Assessment of Subcutaneous Administration of DM199 in Normal Healthy Subjects
Brief Title: An Open Label, Phase 1b, Ascending Dose Study of DM199
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DiaMedica Therapeutics Inc (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DM199-2016-001
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — DM199

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Low dose (Part A) (Experimental): Recombinant human tissue kallikrein
  Interventions: Drug: Recombinant human tissue kallikrein
- Medium low dose (Part A) (Experimental): Recombinant human tissue kallikrein
  Interventions: Drug: Recombinant human tissue kallikrein
- Medium high dose (Part A) (Experimental): Recombinant human tissue kallikrein
  Interventions: Drug: Recombinant human tissue kallikrein
- High dose (Part A) (Experimental): Recombinant human tissue kallikrein
  Interventions: Drug: Recombinant human tissue kallikrein
- Subcutaneous (Part B) (Experimental): Recombinant human tissue kallikrein
  Interventions: Drug: Recombinant human tissue kallikrein
- IV (Part B) (Experimental): Recombinant human tissue kallikrein
  Interventions: Drug: Recombinant human tissue kallikrein

INTERVENTIONS:
Drug: Recombinant human tissue kallikrein — Intravenous DM199
  Other Names: DM199

SUMMARY:
This is a Phase 1B study to assess the safety, tolerability and pharmacokinetics of DM199 in healthy volunteers. The study will be consist of two parts: Part A will focus on intravenous dosing and Part B will directly compare intravenous dosing with subcutaneous dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 50 years of age (inclusive);
2. Healthy with no clinically significant medical problems;
3. BMI between 18 to 30 kg/m2 with a weight between 50 to 100 kg (both inclusive);
4. No history of alcohol or drug abuse (Paracetamol, Barbiturates, Benzodiazepines, Cocaine, Methadone, Amphetamines, Methamphetamines, Opiates, Phencyclidine, Tetrahydrocannabinol (cannabis), Tricyclic Antidepressants). Subjects should be enrolled only after passing the urine drug screen (positive test for paracetamol will be allowed);
5. Non-smokers or light smokers (Less than 5 cigarettes per day) by history and planned during the study;
6. No history of significant allergic diathesis such as urticaria, angioedema or anaphylaxis;
7. Receiving no chronic medications that affect blood pressure control, the bradykinin or angiotensin system including angiotensin-converting-enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB);
8. Willing and able to sign written, informed consent.

Exclusion Criteria:

1. Any significant past or current cardiac, pulmonary, hepatic, renal or other medical condition which in the opinion of the investigator would make participation of the subject in this study medically unsafe or compromise the accuracy of assessment of safety, pharmacokinetic and pharmacodynamic data of the study;
2. Subjects who have abnormal safety labs outside the local lab ranges will be excluded at PI's discretion based on his/her assessment of clinical significance (can be repeated once at screening at PI's discretion);
3. Subjects with past medical history of malignancy except basal cell or squamous cell carcinoma of the skin who have had curative surgical treatment and at least 6 months have elapsed since the procedure;
4. A value outside the specified range of 90 mm Hg - 140 mm Hg for systolic blood pressure and 50 mm Hg - 90 mm Hg for diastolic blood pressure (both inclusive) at screening (can be repeated once at screening as per PI's discretion);
5. Subjects using angiotensin-converting-enzyme inhibitors (ACEi) or angiotensin receptor blockers (ARB) to control blood pressure;
6. History of clinically significant acute bacterial, viral, or fungal systemic infections in the last 4 weeks prior to screening;
7. Clinical or laboratory evidence of an active infection at the time of screening;
8. Known alpha 1-antitrypsin deficiency (α1-antitrypsin deficiency);
9. Serological evidence of human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus (Anti-HCV) at screening;
10. Vaccination within 3 months of screening for the study or requiring vaccination during the study or within 3 months after completion of the study;
11. Females who are pregnant or nursing;
12. Females of childbearing potential (i.e., any woman who is not surgically sterile e.g., hysterectomy, bilateral oophorectomy or >1-year postmenopause status confirmed by follicle-stimulating hormone (FSH) levels as defined by established lab ranges) and all men who, if participating in heterosexual sexual activity that could lead to pregnancy are unable or unwilling to practice medically effective contraception during the study. They should agree to use two reliable methods of contraception (e.g., double-barrier condom plus diaphragm, condom or diaphragm plus a stable dose of hormonal contraception) throughout the study period and until 3 months after receiving study drug. Women of childbearing potential will require compulsory pregnancy testing. A negative pregnancy test (serum and urine) will be documented during screening and at Day -1 respectively;
13. Participation in any other drug study within 8 weeks or 5 half-lives of the study drug, whichever is longer;
14. Unable or unwilling to comply with the protocol requirements for study visits and procedures;
15. Subjects who do not have good venous access for infusion of study drug or for blood sampling;

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days
  Assessment of safety of intravenous dosing

SECONDARY OUTCOMES:
Concentration of DM199 in plasma | 3 days
  Assess plasma drug levels
Concentration of bradykinin in plasma | 3 days
  Assess drug associated biomarkers (e.g. plasma bradykinin levels)

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Perth, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Safety, tolerability and pharmacokinetic profile of recombinant human tissue kallikrein, DM199, after intravenous and subcutaneous administration in healthy volunteers — http://www.ijclinicaltrials.com/index.php/ijct/article/view/238/129